CLINICAL TRIAL: NCT03233204
Title: NCI-COG Pediatric MATCH (Molecular Analysis for Therapy Choice)- A Phase 2 Subprotocol of Olaparib in Patients With Tumors Harboring Defects in DNA Damage Repair Genes
Brief Title: Olaparib in Treating Patients With Relapsed or Refractory Advanced Solid Tumors, Non-Hodgkin Lymphoma, or Histiocytic Disorders With Defects in DNA Damage Repair Genes (A Pediatric MATCH Treatment Trial)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2017-00766; NCI-2017-00766 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); APEC1621H; APEC1621H (Other: Children's Oncology Group); APEC1621H (Other: CTEP); U10CA180886 (NIH)
Record Dates: First submitted 2017-07-25; First posted 2017-07-28 (Actual); Results first posted 2024-04-25 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Advanced Malignant Solid Neoplasm; Ann Arbor Stage III Childhood Non-Hodgkin Lymphoma; Ann Arbor Stage IV Childhood Non-Hodgkin Lymphoma; Low Grade Glioma; Malignant Glioma; Recurrent Childhood Central Nervous System Neoplasm; Recurrent Childhood Ependymoma; Recurrent Childhood Malignant Germ Cell Tumor; Recurrent Childhood Non-Hodgkin Lymphoma; Recurrent Childhood Rhabdomyosarcoma; Recurrent Childhood Soft Tissue Sarcoma; Recurrent Ewing Sarcoma/Peripheral Primitive Neuroectodermal Tumor; Recurrent Glioma; Recurrent Hepatoblastoma; Recurrent Langerhans Cell Histiocytosis; Recurrent Malignant Solid Neoplasm; Recurrent Medulloblastoma; Recurrent Neuroblastoma; Recurrent Osteosarcoma; Refractory Childhood Malignant Germ Cell Tumor; Refractory Ependymoma; Refractory Ewing Sarcoma/Peripheral Primitive Neuroectodermal Tumor; Refractory Glioma; Refractory Hepatoblastoma; Refractory Langerhans Cell Histiocytosis; Refractory Malignant Glioma; Refractory Malignant Solid Neoplasm; Refractory Medulloblastoma; Refractory Neuroblastoma; Refractory Non-Hodgkin Lymphoma; Refractory Osteosarcoma; Refractory Primary Central Nervous System Neoplasm; Refractory Rhabdomyosarcoma; Refractory Soft Tissue Sarcoma; Rhabdoid Tumor; Wilms Tumor
MeSH Terms: conditions — Glioma; Central Nervous System Neoplasms; Familial ependymoma; Neuroectodermal Tumors, Primitive, Peripheral; Hepatoblastoma; Histiocytosis, Langerhans-Cell; Medulloblastoma; Neuroblastoma; Osteosarcoma; Ependymoma; Lymphoma, Non-Hodgkin; Rhabdomyosarcoma; Sarcoma; Rhabdoid Tumor; Wilms Tumor | interventions — olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (olaparib) (Experimental): Patients receive olaparib PO BID on days 1-28. Cycles repeat every 28 days for 2 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Olaparib

INTERVENTIONS:
Drug: Olaparib — Given PO
  Other Names: AZD 2281; AZD-2281; AZD2281; KU 0059436; KU-0059436; KU0059436; Lynparza; Olanib; Olaparix; PARP Inhibitor AZD2281

SUMMARY:
This phase II Pediatric MATCH trial studies how well olaparib works in treating patients with solid tumors, non-Hodgkin lymphoma, or histiocytic disorders with defects in deoxyribonucleic acid (DNA) damage repair genes that have spread to other places in the body (advanced) and have come back (relapsed) or do not respond to treatment (refractory). Olaparib is an inhibitor of PARP, an enzyme that helps repair DNA when it becomes damaged. Blocking PARP may help keep cancer cells from repairing their damaged DNA, causing them to die. PARP inhibitors are a type of targeted therapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the objective response rate (ORR; complete response + partial response) in pediatric patients treated with olaparib with advanced solid tumors (including central nervous system [CNS] tumors), non-Hodgkin lymphomas or histiocytic disorders that harbor activating genetic alterations in the deleterious genetic alterations in the DNA damage repair (DDR) pathway.

SECONDARY OBJECTIVES:

I. To estimate the progression free survival in pediatric patients treated with olaparib with advanced solid tumors including non-Hodgkin lymphomas, CNS tumors, and histiocytosis that harbor deleterious genetic alterations in the DDR pathway.

II. To obtain information about the tolerability of olaparib in children and adolescents with relapsed or refractory cancer.

III. To provide preliminary estimates of the pharmacokinetics of olaparib in children and adolescents with relapsed or refractory cancer.

EXPLORATORY OBJECTIVE:

I. To explore approaches to profiling changes in tumor genomics over time through the evaluation of circulating tumor DNA.

OUTLINE:

Patients receive olaparib orally (PO) twice daily (BID) on days 1-28. Cycles repeat every 28 days for 2 years in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have enrolled onto APEC1621SC (NCT03155620) and must have been given a treatment assignment to Molecular Analysis for Therapy Choice (MATCH) to APEC1621H based on the presence of an actionable mutation
* Patients must be >= than 12 months and =< 21 years of age at the time of study enrollment
* Patients must have a body surface area >= 0.65 m^2 at enrollment
* Patients must have radiographically measurable disease at the time of study enrollment; patients with neuroblastoma who do not have measurable disease but have iobenguane (MIBG) positive (+) evaluable disease are eligible; measurable disease in patients with CNS involvement is defined as tumor that is measurable in two perpendicular diameters on magnetic resonance imaging (MRI) and visible on more than one slice

  * Note: The following do not qualify as measurable disease:

    * Malignant fluid collections (e.g., ascites, pleural effusions)
    * Bone marrow infiltration except that detected by MIBG scan for neuroblastoma
    * Lesions only detected by nuclear medicine studies (e.g., bone, gallium or positron emission tomography [PET] scans) except as noted for neuroblastoma
    * Elevated tumor markers in plasma or cerebrospinal fluid (CSF)
    * Previously radiated lesions that have not demonstrated clear progression post radiation
    * Leptomeningeal lesions that do not meet the measurement requirements for Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
* Karnofsky >= 50% for patients > 16 years of age and Lansky >= 50 for patients =< 16 years of age

  * Note: Neurologic deficits in patients with CNS tumors must have been relatively stable for at least 7 days prior to study enrollment; patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score
* Patients must have fully recovered from the acute toxic effects of all prior anti-cancer therapy and must meet the following minimum duration from prior anti-cancer directed therapy prior to enrollment; if after the required timeframe, the numerical eligibility criteria are met, e.g. blood count criteria, the patient is considered to have recovered adequately

  * Cytotoxic chemotherapy or other anti-cancer agents known to be myelosuppressive

    * >= 21 days after the last dose of cytotoxic or myelosuppressive chemotherapy (42 days if prior nitrosourea)
  * Anti-cancer agents not known to be myelosuppressive (e.g. not associated with reduced platelet or absolute neutrophil count [ANC] counts): >= 7 days after the last dose of agent
  * Antibodies: >= 21 days must have elapsed from infusion of last dose of antibody, and toxicity related to prior antibody therapy must be recovered to grade =< 1
  * Corticosteroids: If used to modify immune adverse events related to prior therapy, >= 14 days must have elapsed since last dose of corticosteroid
  * Hematopoietic growth factors: >= 14 days after the last dose of a long-acting growth factor (e.g. pegfilgrastim) or 7 days for short-acting growth factor; for growth factors that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur; the duration of this interval must be discussed with the study chair and the study-assigned research coordinator
  * Interleukins, interferons and cytokines (other than hematopoietic growth factors): >= 21 days after the completion of interleukins, interferon or cytokines (other than hematopoietic growth factors)
  * Stem cell infusions (with or without total body irradiation [TBI]):

    * Allogeneic (non-autologous) bone marrow or stem cell transplant, or any stem cell infusion including donor lymphocyte infusion (DLI) or boost infusion: >= 84 days after infusion and no evidence of graft versus host disease (GVHD)
    * Autologous stem cell infusion including boost infusion: >= 42 days
  * Cellular therapy: >= 42 days after the completion of any type of cellular therapy (e.g. modified T cells, natural killer [NK] cells, dendritic cells, etc.)
  * Radiation therapy (XRT)/external beam irradiation including protons: >= 14 days after local XRT; >= 150 days after TBI, craniospinal XRT or if radiation to >= 50% of the pelvis; >= 42 days if other substantial bone marrow (BM) radiation

    * Note: Radiation may not be delivered to "measurable disease" tumor site(s) being used to follow response to subprotocol treatment
  * Radiopharmaceutical therapy (e.g., radiolabeled antibody, 131iodine [I]-MIBG): >= 42 days after systemically administered radiopharmaceutical therapy
  * Patients must not have received prior exposure to olaparib, veliparib, niraparib, rucaparib, talazoparib or other poly adenosine diphosphate ribose polymerase inhibitors (PARPi)
* For patients with solid tumors without known bone marrow involvement: peripheral absolute neutrophil count (ANC) >= 1000/mm^3 (within 7 days prior to enrollment)
* For patients with solid tumors without known bone marrow involvement: platelet count >= 100,000/mm^3 (within 7 days prior to enrollment) (transfusion independent, defined as not receiving platelet transfusions for at least 7 days prior to enrollment)
* Patients with known bone marrow metastatic disease will be eligible for study provided they meet the blood counts (may receive platelet or packed red blood cells [pRBC] transfusions provided they are not known to be refractory to red cell or platelet transfusions); these patients will not be evaluable for hematologic toxicity
* Creatinine clearance or radioisotope glomerular filtration rate (GFR) >= 70 ml/min/1.73 m^2 (within 7 days prior to enrollment) or
* A serum creatinine based on age/gender as follows (within 7 days prior to enrollment):

  * Age 1 to < 2 years: maximum serum creatinine 0.6 mg/dL for male and 0.6 mg/dL for female
  * Age 2 to < 6 years: maximum serum creatinine 0.8 mg/dL for male and 0.8 mg/dL for female
  * Age 6 to < 10 years: maximum serum creatinine 1 mg/dL for male and 1 mg/dL for female
  * Age 10 to < 13 years: maximum serum creatinine 1.2 mg/dL for male and 1.2 mg/dL for female
  * Age 13 to < 16 years: maximum serum creatinine 1.5 mg/dL for male and 1.4 mg/dL for female
  * Age >= 16 years: maximum serum creatinine 1.7 mg/dL for male and 1.4 mg/dL for female
* Patients with solid tumors: bilirubin (sum of conjugated + unconjugated) =< 1.5 x upper limit of normal (ULN) for age (within 7 days prior to enrollment)
* Patients with solid tumors: serum glutamic pyruvic transaminase (SGPT) (alanine aminotransferase [ALT]) =< 135 U/L (within 7 days prior to enrollment); (for the purpose of this study, the ULN for SGPT is 45 U/L)
* Patients with solid tumors: serum albumin >= 2 g/dL (within 7 days prior to enrollment)
* Activated partial thromboplastin time (aPTT) =< 1.5 x ULN (within 7 days prior to enrollment)
* International normalized ratio (INR) =< 1.5 (within 7 days prior to enrollment)
* Patients must be able to swallow intact tablets
* All patients and/or their parents or legally authorized representatives must sign a written informed consent; assent, when appropriate, will be obtained according to institutional guidelines

Exclusion Criteria:

* Pregnant or breast-feeding women will not be entered on this study due to risks of fetal and teratogenic adverse events as seen in animal/human studies; pregnancy tests must be obtained in girls who are post-menarchal; women of child-bearing potential and their partners should agree to use two (2) highly effective forms of contraception throughout study participation and for at least one (1) month after the last dose of olaparib; male study participants should avoid fathering a child or donating sperm during the study and for three (3) months after the last dose of olaparib
* Concomitant medications

  * Corticosteroids: patients receiving corticosteroids who have not been on a stable or decreasing dose of corticosteroid for at least 7 days prior to enrollment are not eligible; if used to modify immune adverse events related to prior therapy, >= 14 days must have elapsed since last dose of corticosteroid
  * Investigational drugs: patients who are currently receiving another investigational drug are not eligible
  * Anti-cancer agents: patients who are currently receiving other anti-cancer agents are not eligible
  * Anti-GVHD agents post-transplant: patients who are receiving cyclosporine, tacrolimus or other agents to prevent graft-versus-host disease post bone marrow transplant are not eligible for this trial
  * CYP3A/CYP3A4 agents: patients who are currently receiving drugs that are strong and moderate inducers or inhibitors of CYP3A or CYP3A4 are not eligible; strong inducers or inhibitors of CYP3A4 should be avoided from 21 days prior to enrollment to the end of the study
* Patients who have an uncontrolled infection are not eligible
* Patient who are known to be serologically positive for human immunodeficiency virus (HIV)
* Patients with known active hepatitis (i.e. hepatitis B or C)
* Patients who have received a prior solid organ transplantation are not eligible
* Patients with symptomatic uncontrolled brain metastases; a scan to confirm the absence of brain metastases is not required; the patient can receive a stable dose of corticosteroids before and during the study as long as these were started at least 4 weeks prior to enrollment; patients with spinal cord compression unless considered to have received definitive treatment for this and evidence of clinically stable disease for 28 days
* Patients with known symptomatic Fanconi anemia (FA), ataxia-telangiectasia (A-T) syndrome, Bloom syndrome (BS) and Nijmegen breakage syndrome (NBS) are not eligible (asymptomatic carriers are acceptable)
* Major surgery must not have occurred within 2 weeks prior to enrollment and patients must have recovered from any effects of any major surgery
* Patients who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study are not eligible

Ages: 12 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 6 (Actual)
Dates: Start 2017-09-14 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2024-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julia Glade-Bender, Principal Investigator — Children's Oncology Group
Locations (113):
- United States (111):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Banner Children's at Desert, Mesa, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Kaiser Permanente Downey Medical Center, Downey, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Miller Children's and Women's Hospital Long Beach, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Rocky Mountain Hospital for Children-Presbyterian Saint Luke's Medical Center, Denver, Colorado
  - Yale University, New Haven, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Florida Health Science Center - Gainesville, Gainesville, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Children's Healthcare of Atlanta - Egleston, Atlanta, Georgia
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Norton Children's Hospital, Louisville, Kentucky
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Albany Medical Center, Albany, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - NYU Langone Hospital - Long Island, Mineola, New York
  - The Steven and Alexandra Cohen Children's Medical Center of New York, New Hyde Park, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - New York Medical College, Valhalla, New York
  - Mission Hospital, Asheville, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Legacy Emanuel Children's Hospital, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Children's Hospital of San Antonio, San Antonio, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - West Virginia University Healthcare, Morgantown, West Virginia
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Puerto Rico (2):
  - San Jorge Children's Hospital, San Juan
  - University Pediatric Hospital, San Juan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Glade Bender JL, Pinkney K, Williams PM, Roy-Chowdhuri S, Patton DR, Coffey BD, Reid JM, Piao J, Saguilig L, Alonzo TA, Berg SL, Ramirez NC, Fox E, Weigel BJ, Hawkins DS, Mooney MM, Takebe N, Tricoli JV, Janeway KA, Seibel NL, Parsons DW. Olaparib for childhood tumors harboring defects in DNA damage repair genes: arm H of the NCI-COG Pediatric MATCH trial. Oncologist. 2024 Jul 5;29(7):638-e952. doi: 10.1093/oncolo/oyae096. PMID 38815151
- [Derived] Hattinger CM, Patrizio MP, Magagnoli F, Luppi S, Serra M. An update on emerging drugs in osteosarcoma: towards tailored therapies? Expert Opin Emerg Drugs. 2019 Sep;24(3):153-171. doi: 10.1080/14728214.2019.1654455. Epub 2019 Aug 14. PMID 31401903

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Olaparib)
Started | 6
Completed | 0
Not Completed | 6
Not completed — Adverse Event | 1
Not completed — Death | 1
Not completed — Withdrawal by Subject | 1
Not completed — Progressive Disease | 3

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Olaparib)
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 5
  Between 18 and 65 years | 1
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.5 (4.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (Complete Response/Partial Response)
Description: A responder is defined as a patient who achieves a best response of partial response or complete response on the study. Response rates will be calculated as the percent of evaluable patients who are responders, and confidence intervals will be constructed using the Wilson score interval method. The revised Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1) was used to determine response and progression in this study, with specific criteria outlined for the different subtypes of tumors (e.g., 2-dimensional measurements for central nervous system (CNS) tumors).
Time Frame: Up to 2 years from study entry
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Olaparib)
Number analyzed (Participants) | 6
percentage of participants | 0 [0 to 0]

2. Secondary Outcome: Progression Free Survival (PFS)
Description: The Kaplan-Meier method will be used to estimate the 6 month PFS. PFS is defined as time from initiation of protocol treatment to disease progression, recurrence, death from any cause, or date of last contact.
Time Frame: Up to 6 months from study entry
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Olaparib)
Number analyzed (Participants) | 6
percentage of participants | 33.3 [4.6 to 67.6]

3. Secondary Outcome: Percentage of Patients Experiencing Treatment-related Grade 3 or Higher Adverse Events
Description: Percentage of patients experiencing treatment-related grade 3 or higher adverse events will be evaluated according to National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0.
Time Frame: Up to 2 years from study entry
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Olaparib)
Number analyzed (Participants) | 6
percentage of participants | 16.7 [0.4 to 64.1]

4. Secondary Outcome: Pharmacokinetics (PK) of Olaparib, Area Under the Curve (AUC)
Description: The mean (sd) of the AUC.
Time Frame: Up to day 8 of cycle 1
Population: 3 of the 6 enrolled patients had PK data available for analysis
Measure: Mean (Standard Deviation); unit: mcg*hr/ml
Arm/Group | Treatment (Olaparib)
Number analyzed (Participants) | 3
mcg*hr/ml | 48.8 (27.8)

5. Other Pre Specified Outcome: Change in Tumor Genomic Profile
Description: Approaches to profiling changes in tumor genomics over time through evaluation of circulating tumor deoxyribonucleic acid will be explored. Descriptive analysis will be performed and will be summarized with simple summary statistics.
Time Frame: Cycle 5 day 1 to 4 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse Events monitored/assessed from enrollment to 30 days after the end of treatment, up to 2 years. All-Cause Mortality monitored/assessed up to 5 years
Description: Adverse event reporting is collected routinely using case report forms. The SAE table reflects NCI Common Terminology Criteria for Adverse Events (CTCAEs) submitted by the institution via expedited reporting (NCI AdEERs / CAeRs). All remaining CTCAEs collected by means other than expedited reporting are non-serious and are reported in the "AE Other" table. Ineligible patients are excluded from reporting of adverse events. All-Cause Mortality includes all deaths collected on the study.
Arm/Group | Treatment (Olaparib)
All-Cause Mortality (participants affected / at risk) | 4/6
Serious Adverse Events (participants affected / at risk) | 3/6
Other Adverse Events (participants affected / at risk) | 5/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Olaparib) (N=6)
Disease progression (General disorders) | 1
Allergic reaction (Immune system disorders) | 1
Hypercalcemia (Metabolism and nutrition disorders) | 1
Seizure (Nervous system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Olaparib) (N=6)
Anemia (Blood and lymphatic system disorders) | 3
Cardiac disorders - Other, specify (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Eye pain (Eye disorders) | 1
Optic nerve disorder (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 2
Edema limbs (General disorders) | 1
Fatigue (General disorders) | 1
Gait disturbance (General disorders) | 1
General disorders and administration site conditions - Other, specify (General disorders) | 1
Malaise (General disorders) | 1
Conjunctivitis (Infections and infestations) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Creatinine increased (Investigations) | 1
Investigations - Other, specify (Investigations) | 1
Lymphocyte count decreased (Investigations) | 4
Neutrophil count decreased (Investigations) | 1
Platelet count decreased (Investigations) | 1
Weight loss (Investigations) | 1
White blood cell decreased (Investigations) | 3
Anorexia (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hypernatremia (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 2
Dysgeusia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 2
Anxiety (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1
Hematuria (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 2
Hypotension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-09): https://cdn.clinicaltrials.gov/large-docs/04/NCT03233204/Prot_SAP_000.pdf